CLINICAL TRIAL: NCT02612675
Title: Plasma Glucose and Insulin Response to Two Oral Nutrition Supplements in Persons With Type 2 Diabetes Mellitus
Brief Title: Glycemic Response to Oral Nutrition Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13.10.US.HCN
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard ONS (Active Comparator): Nutritional beverage (Oral Nutrition Supplement) designed for oral consumption
  Interventions: Other: ONS
- Low Carbohydrate ONS (Experimental): Nutritional beverage (Oral Nutrition Supplement) designed for oral consumption
  Interventions: Other: ONS

INTERVENTIONS:
Other: ONS

SUMMARY:
This will be a randomized, cross-over study of two oral nutrition supplements in individuals with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 yrs
* Type 2 diabetes controlled with diet or diet and oral agent, with the exception of sulfonylureas such as glimepiride (Amaryl), glipizide (Glucotrol/Glucotrol XL) and glyburide (DiaBeta, Micronase, Glynase Prestabs); meglitinides such as reaglinide (Prandin) and nateglinide (Starlix); and alpha-glucosidase inhibitors such as acarbose (Precose) and miglitol (Glyset)
* Hemoglobin A1C less than 9.0%
* Fasting blood glucose less than 180 mg

Exclusion Criteria:

* Allergy to milk protein or any other component of the formula

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Area under the blood glucose curve (AUC 0-240) | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sherwyn Schwartz, MD, Principal Investigator — Diabetes & Glandular Disease Clinic, PA
Locations (1):
- Diabetes & Glandular Disease Clinic, PA, San Antonio, Texas, United States

REFERENCES:
- [Derived] Huhmann MB, Smith KN, Schwartz SL, Haller SK, Irvin S, Cohen SS. Plasma glucose and insulin response to two oral nutrition supplements in adults with type 2 diabetes mellitus. BMJ Open Diabetes Res Care. 2016 Aug 31;4(1):e000240. doi: 10.1136/bmjdrc-2016-000240. eCollection 2016. PMID 27648290